CLINICAL TRIAL: NCT00177346
Title: A Randomized Trial of Carotid Artery Stenting With and Without Cerebral Protection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MakarounIDE; 0
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis

ARMS (2):
- CAS with cerebral protection (Experimental)
  Interventions: Device: CAS with cerebral protection
- CAS without cerebral protection (Active Comparator)
  Interventions: Device: CAS without cerebral protection

INTERVENTIONS:
Device: CAS with cerebral protection
  Arms: CAS with cerebral protection
Device: CAS without cerebral protection
  Arms: CAS without cerebral protection

SUMMARY:
The primary objective of this study is to evaluate carotid artery stenting (CAS) with and without cerebral protection (CP) to determine if CP improves safety and effectiveness of CAS.

DETAILED DESCRIPTION:
This study is a single center, prospective, randomized trial evaluating the safety and effectiveness of CAS with and without CP. The study population will be comprised of subjects with atherosclerotic, post endarterectomy restenotic or other obstructive lesions in native carotid arteries. Other carotid artery pathology not amenable to surgical repair (for example carotid artery dissection) will also be considered. Subjects at high risk for complications from standard CEA will be the target population for this study. High risk status will be confirmed by two physicians, one of whom is a vascular surgeon. Both symptomatic and asymptomatic subjects will be enrolled. This will ensure that the proportion of symptomatic subjects is the same in the two arms of the study. "Symptomatic" is defined in the exclusion criteria. The expected duration of this clinical trial is 3 years.

In this study there are there are two arms that a subject may be randomized to:

Group1: CAS with the use of the RX ACCUNET Group 2: CAS without the use of the RX ACCUNET This study has been designed to test whether the addition of CP enhances the safety and effectiveness of CAS.

ELIGIBILITY:
Inclusion Criteria:

* To participate in this study, the subject MUST have all of the following for inclusion in the study:

  • The subject (male or non-pregnant female) must be > 18 years of age.

  • The subject should have a stenosis in the common or internal carotid artery of at least 70% determined by one of the modalities listed below.

  • The subject should be considered a relatively high risk for carotid endarterectomy. This determination has to be made and documented by two physicians, at least one of who must be a vascular surgeon acting as an investigator on this trial. High risk considerations should include at least one of the following:
  1. Cardiac dysfunction. NYHA class III or above, compensated or active congestive heart failure (CHF), incomplete coronary revascularization, ejection fraction of <35%, pulmonary hypertension, or recommendation of a cardiologist against open CEA.
  2. Pulmonary dysfunction, history of respiratory failure, severe chronic obstructive pulmonary Disease (COPD) on bronchodilators or recommendation of a pulmonary specialist against open CEA.
  3. Multi-system dysfunction, defined as any combination of medical problems in three distinct systems.
  4. Anatomic issues: previous CEA or neck dissection, neck irradiation, inaccessible lesions, neck fusion or other anatomic considerations increasing the risk of CEA.
  5. Age >80 AND symptomatic (defined below)
  6. General debilitation documented by the subject's primary physician.
  7. Increased anesthetic risk as documented by an anesthesiologist.

     * Subjects can be either clinically symptomatic or asymptomatic (less than 80 years of age). Symptomatic subjects will have experienced an event within the previous 120 days in the ipsilateral carotid artery distribution. The event will be classified as either 1) one or more TIAs, characterized by distinct focal neurologic dysfunction or monocular blindness with clearing of signs and symptoms within 24 hours, or 2) one or more completed strokes (as defined by this protocol) with persistence of symptoms or signs for more than 24 hours (the most recent event is used as the qualifying event).

       **Patients with major non-hemorrhagic strokes will be included if their clinical status has been stable for 5 days (based on an exam performed by a neurologist participating as a Co-Investigator in this trial).
     * If an angiogram is performed to qualify the subject, it should be as recent as feasible and will not be acceptable if done > 120 days from study entry. Angiograms from other institutions will be acceptable.
     * Other non-invasive qualifying imaging modalities include:

  <!-- -->

  1. Duplex ultrasound (DU) performed at UPMC Presbyterian or Shadyside hospitals.
  2. Magnetic Resonance Angiography (MRA) performed at UPMC Presbyterian or Shadyside hospitals.
  3. Computed Tomographic Angiography (CTA) performed at UPMC Presbyterian or Shadyside hospitals.

     * The degree of stenosis from these non-invasive studies has to be confirmed on the pre-deployment diagnostic angiography prior to proceeding with stent deployment.
     * However, if two of the non-invasive studies listed above report a stenosis of >70%, AND the pre-deployment angiogram reveals a 50 -70% stenosis, the patient will be randomized and entered into the trial as the angiogram can on occasion underestimate the stenosis.

       * Female subjects of childbearing potential must have a documented negative pregnancy test during the index hospitalization.
       * The subject must sign a written informed consent, prior to the procedure, using a form that is approved by the local Institutional Review Board or Medical Ethics Committee.
       * If a patient's creatinine is 3.5 or greater, their nephrologist must clear them to participate in the trial.

     Exclusion Criteria:
* To participate in this study, the subject may NOT HAVE any of the following at enrollment to the study:

  * The subject has had an intracranial hemorrhage, hemorrhagic stroke, or any stroke with mass effect demonstrated on CT scan or MRI within 30 days of the index procedure.
  * The subject has a persisting ischemic stroke (defined as either a score > 15 on the NIH stroke scale, a Rankin score > 3 or a Barthel score < 60 measured within one week prior to study entry).
  * The subject has an intracranial mass lesion (i.e., abscess, tumor, or other infection).
  * The subject has known allergies to heparin, to both ticlopidine and clopidogrel or to metals used in stents.
  * There is any visual angiographic evidence of intraluminal thrombus thought to increase the risk of plaque fragmentation and distal embolization.
  * The subject has peripheral vascular, supra-aortic or internal carotid artery tortuosity precluding use of catheter-based techniques required for successful results.
  * The subject, if female, has a positive pregnancy test.
  * The subject has an arterio-venous malformation in the territory of the target carotid artery.
  * Subjects with highly calcified lesions resistant to predilation by PTA
  * The subject has unstable angina (defined as Class IV or at rest), evolving MI or recent MI (within 14 days).
  * The subject has any condition that precludes adequate local hemostasis.
  * Patients who are not candidates for MRI scanning (pacemaker, etc).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint
Safety: The 30-day composite of stroke or death,
Effectiveness: The percentage of subjects who show evidence of new ischemic injury on diffusion MRI imaging, as well as the amount of infarcted tissue

SECONDARY OUTCOMES:
Secondary Endpoints
Successful stent deployment at the target lesion,
Successful CP device deployment and retrieval,
Successful resolution of the stenosis (<30% residual stenosis) determined by angiography immediately post-stent placement,
Access site vascular complications, defined as need for surgical repair or blood transfusion,
Restenosis (>50% diameter reduction) rates both in-stent or of the adjacent artery determined by carotid ultrasound imaging at 1 year post-procedure,
Ipsilateral neurologic deficits on neurologic assessments at 24 hours and 30 days post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Michel S Makaroun, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center Presbyterian &Shadyside Hospitals, Pittsburgh, Pennsylvania, United States